CLINICAL TRIAL: NCT01971307
Title: Supporting Primary Care in Diagnosis and Choice of Treatment for Patients With Psychosocial Symptoms: SGEPsyScan.
Acronym: SGE-PsyScan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Stichting Gezondheidscentra Eindhoven (SGE) (Unknown); Stichting Volksgezondheidszorg (VGZ) (Unknown); Zorgverzekeraar CZ (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: NL44597.068.13/ METC 13-3-034
Record Dates: First submitted 2013-10-11; First posted 2013-10-29 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Mental Disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SGE-PsyScan (Experimental): The SGE-PsyScan is an internet application to which the General Practitioner (GP) refers the patient, which includes the distress screener, the 4-Dimensional Symptom Questionnaire (4DSQ) and a series of additional questions for differentiating between stress, depressive, anxious and somatization symptoms. Based on the 4DSQ patients and GPs receive advices for possible treatments.
  Interventions: Other: SGE-PsyScan
- Usual care (No Intervention): Usual care for persons with psychosocial symptoms and disorders in Dutch primary care includes all usual care procedures; preventive, screening, diagnostic, (non-)pharmacological or therapeutic procedures which are routinely used in everyday care.

INTERVENTIONS:
Other: SGE-PsyScan
  Arms: SGE-PsyScan

SUMMARY:
Although effective treatments for psychosocial symptoms and disorders are available, patients frequently do not receive the most appropriate and effective treatment for their symptoms because of inappropriate and unstructured diagnostics of psychosocial symptoms in general practice. The hypothesis is that by using the intervention SGE-PsyScan the clinical symptoms of patients can be assessed more uniformly and earlier as opposed to the GPs' assessment in usual care. As a result, patients are supposed to start earlier with a treatment that fits the type and severity of their symptoms better.

The patients will be randomly assigned to either receive the SGE-PsyScan or usual care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with (suspected) psychosocial symptoms
* Aged 18 years or older and capacitated
* Adequate understanding of Dutch language
* Able to perform SGE-PsyScan at home, individually

Exclusion Criteria:

* Clear and treatable somatic causes of symptoms
* Acute distress/danger
* No written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2013-12; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
The rate of patients who achieve a successful decrease in the level of psychosocial symptoms as measured with the Symptom Checklist 90 (SCL-90) after 12 months. A successful treatment result is defined as a decrease in the SCL-90 patient score of 50%. | 12 months

SECONDARY OUTCOMES:
The level of psychosocial symptoms of patients as measured with the SCL-90 | 3 months
The level of psychosocial symptoms of patients as measured with the SCL-90 | 6 months
Health technology assessment | 3 months
  We will measure direct and indirect costs in both groups with the Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness (TiC-P) and Electronic Medical Records (EMR) parameters indicating relevant expenditures including treatments, consultations and referrals
Health technology assessment | 6 months
  We will measure direct and indirect costs in both groups with the Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness (TiC-P) and Electronic Medical Records (EMR) parameters indicating relevant expenditures including treatments, consultations and referrals
Health technology assessment | 9 months
  We will measure direct and indirect costs in both groups with the Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness (TiC-P) and Electronic Medical Records (EMR) parameters indicating relevant expenditures including treatments, consultations and referrals
Health technology assessment | 12 months
  We will measure direct and indirect costs in both groups with the Trimbos/iMTA questionnaire for Costs associated with Psychiatric Illness (TiC-P) and Electronic Medical Records (EMR) parameters indicating relevant expenditures including treatments, consultations and referrals
Quality of life will be measured using the EuroQol-5Dimensions-5Levels (EQ-5D-5L) questionnaire | 3 months
Quality of life will be measured using the EuroQol-5Dimensions-5Levels (EQ-5D-5L) questionnaire | 6 months
Quality of life will be measured using the EuroQol-5Dimensions-5Levels (EQ-5D-5L) questionnaire | 12 months
The extent of patient satisfaction with the care they receive, will be measured using the Patient Assessment of Chronic Illness Care (PACIC) | 3 months
The extent of patient satisfaction with the care they receive, will be measured using the Patient Assessment of Chronic Illness Care (PACIC) | 6 months
The extent of patient satisfaction with the care they receive, will be measured using the Patient Assessment of Chronic Illness Care (PACIC) | 12 months
Electronic medical records parameters | 12 months
  Relevant psychosocial care parameters will be extracted from the EMR to monitor changes in care patterns including previous psychosocial episodes, numbers and types of psychosocial diagnoses, use of screening/diagnostic instruments, comorbidity, treatments, medication prescriptions, referrals and health care consumption.

OTHER OUTCOMES:
Health care provider satisfaction with the Assessment of Chronic Illness Care (ACIC) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Mark G Spigt, PhD, Principal Investigator — Research Institute CAPHRI, Department of Family Medicine, Maastricht University
Locations (1):
- Stichting Gezondheidscentra Eindhoven, Eindhoven, Netherlands

REFERENCES:
- [Derived] Gidding LG, Spigt M, Winkens B, Herijgers O, Dinant GJ. PsyScan e-tool to support diagnosis and management of psychological problems in general practice: a randomised controlled trial. Br J Gen Pract. 2018 Jan;68(666):e18-e27. doi: 10.3399/bjgp17X694109. Epub 2017 Dec 18. PMID 29255109